CLINICAL TRIAL: NCT00437567
Title: Prebiotics vs. Placebo in the Prevention of Necrotizing Enterocolitis in Premature Neonates
Brief Title: Prebiotics in the Prevention of Necrotizing Enterocolitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Cathy Hammerman, Professor of Pediatrics, Shaare Zedek Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SZMC/CH/32007
Record Dates: First submitted 2007-02-08; First posted 2007-02-21 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Necrotizing Enterocolitis
Keywords: galacto-oligosaccharides; prebiotics; NEC
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — 4'-galactooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prebiotics (Active Comparator): Babies randomized to this arm will receive galacto-oligosaccharide supplements
  Interventions: Dietary Supplement: Galacto-oligosaccharide (GOS)
- Placebo (Placebo Comparator): Babies randomized to this arm will receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Galacto-oligosaccharide (GOS) — Treatment group to receive 1.3 gm/kg/day GOS from initiation of enteral feeds until 35 weeks post-conceptual age.
  Arms: Prebiotics
Other: Placebo — Similar quantity of sterile water to be added to milk
  Arms: Placebo

SUMMARY:
Necrotizing enterocolitis (NEC) is the most common gastrointestinal catastrophe affecting 10-15% of premature neonates of <1500 gm. NEC is a disease of the immature intestine, characterized by impaired mucosal barrier function leading to increased gut permeability. We have previously demonstrated a protective effect of probiotic administration against the development of NEC. Others have shown that prebiotics can stimulate natural production of bifidobacteria and lactobacillus in the preterm gut. We have therefore hypothesized that prophylactic administration of prebiotics would also provide protection against necrotizing enterocolitis in the premature neonate, without the potential for sepsis which has been reported on rare occasions with probiotics administration.

DETAILED DESCRIPTION:
Specifically, we hope to demonstrate that fewer of the babies who are treated with galacto-oligosaccharides (GOS) will develop NEC as compared with controls.

Preterm neonates, <1750 gm birth weight will potentially be candidates for study. They will be randomly assigned to receive one of two milk additives from the time enteral feeds are begun until 35 weeks post-conceptual age: prebiotics (GOS) or placebo (water). All infants will be followed prospectively for signs of feeding intolerance and/or development of NEC. These will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates
* < 1750 gm birth weight

Exclusion Criteria:

* Infants who are deemed unlikely to survive
* Infants with significant congenital malformations
* Infants with other gastrointestinal problems

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Necrotizing Enterocolitis | yearly

SECONDARY OUTCOMES:
fecal calprotectin, urine IFABP | end of study
NEC related morbidity, ie. perforation, surgery [including peritoneal drain placement] | yearly
Stool bifidobacteria | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Hammerman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Bin-Nun A, Bromiker R, Wilschanski M, Kaplan M, Rudensky B, Caplan M, Hammerman C. Oral probiotics prevent necrotizing enterocolitis in very low birth weight neonates. J Pediatr. 2005 Aug;147(2):192-6. doi: 10.1016/j.jpeds.2005.03.054. PMID 16126048